CLINICAL TRIAL: NCT04426006
Title: Serological Response to SARS-Cov-2 Virus in Personnel of the Institut Bergonié in the Context of the COVID-19 Pandemic - PRO-SERO-COV
Brief Title: Serological Response to SARS-Cov-2 Virus in Personnel of the Institut Bergonié in the Context of the COVID-19 Pandemic
Acronym: PRO-SERO-COV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IB 2020-01; 2020-A01355-34 (Other: ANSM ID-RCB number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2023-04

CONDITIONS: Sars-CoV2; Serum; Disease
Keywords: COVID-19; Health professionals; Serology; SARS-CoV-2 Antibodies; Anxiety; ELISA
MeSH Terms: conditions — Disease; COVID-19; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO-SERO-COV (Other): Blood sample and self-administered questionnaire
  Interventions: Other: PRO-SERO-COV

INTERVENTIONS:
Other: PRO-SERO-COV — At inclusion, 3 months and 12 months :
  * blood sample (2 x 5ml)
  * self-administered questionnaire

SUMMARY:
The question of the immune response of the population, particularly of professional populations in contact with vulnerable populations (such as those with chronic conditions such as cancer), is an important issue. Knowing the evolution of this response over time in this population can help answer outstanding questions. The PRO-SERO-COV study is a seroprevalence study of caregivers working in the hospital sector with a follow-up at 3 months and 12 months. The objective is to evaluate and monitor at 3 and 12 months the serological immune status to an infection by the SARS-CoV-2 virus in active volunteer professionals working at the Institut Bergonié with different types of exposure: healthcare professionals and professionals in other services.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years-old and older.
2. Person in employment (on fixed-term or permanent contracts) since (at least) March 17th, 2020, the date of national implementation of containment measures in response to the COVID-19 pandemic.
3. Signed informed consent.
4. Person affiliated to a French social security regimen in accordance with Article 1121-11 of the French Public Health Code).

Exclusion Criteria:

1. Report of known active SARS-CoV-2 infection within 10 days prior to the date of signing the consent. Known active SARS-CoV-2 infection is defined as a positive result on a diagnostic RT-PCR test.
2. Presence of known symptoms suggestive of COVID-19 within 10 days prior to the date of signing consent: fever, fatigue, dry cough, shortness of breath, loss of taste and/or smell, headache, body aches, aches and pains, conjunctivitis or colds, digestive disorders (vomiting, diarrhea).
3. A person who is unable to follow and comply with research procedures due to geographical, social or psychological reasons.
4. Pregnant or breastfeeding woman.
5. Person deprived of their liberty, incapable or incapable of giving their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone MATHOULIN-PELISSIER, MD, PhD, Study Chair — s.mathoulin@bordeaux.unicancer.fr
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richez B, Cantarel C, Durrieu F, Soubeyran I, Blanchi J, Pernot S, Chakiba Brugere C, Roubaud G, Cousin S, Etienne G, Floquet A, Babre F, Rivalan J, Lalet C, Narbonne M, Belaroussi Y, Bellera C, Mathoulin-Pelissier S. One-Year Follow-Up of Seroprevalence of SARS-CoV-2 Infection and Anxiety among Health Workers of a French Cancer Center: The PRO-SERO-COV Study. Int J Environ Res Public Health. 2023 May 25;20(11):5949. doi: 10.3390/ijerph20115949. PMID 37297553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusions from June 18th, 2020 to September 28th, 2020 in the Institut Bergonié (Bordeaux, France)
Groups:
- PRO-SERO-COV: Blood sample and self-administered questionnaire
  PRO-SERO-COV: At inclusion, 3 months and 12 months :
  * blood sample (2 x 5ml)
  * self-administered questionnaire
Period: Inclusion
Arm/Group | PRO-SERO-COV
Started | 526
Completed (Participants who completed the self-administered questionnaire and had blood sample at inclusion) | 517
Not Completed | 9
Not completed — Protocol Violation | 1
Not completed — Self-administered questionnaire at inclusion not completed | 7
Not completed — Blood sample at inclusion not done | 1
Period: 3 Months
Arm/Group | PRO-SERO-COV
Started | 517
Completed | 500
Not Completed | 17
Not completed — Lost to Follow-up | 17
Period: 12 Months
Arm/Group | PRO-SERO-COV
Started | 500
Completed | 462
Not Completed | 38
Not completed — Lost to Follow-up | 38

BASELINE CHARACTERISTICS:
Arm/Group | PRO-SERO-COV
Number analyzed (Participants) | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 431
  Male | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Positive Serological Immune Status to a Previous Infection by the SARS-CoV-2 Virus at Inclusion
Description: Total antibodies (IgG and IgM) directed against the N (nucleocapsid) protein of the virus were determined by ECLIA on a Cobas® 8000 (Roche Diagnostic, France) with the Elecsys Anti-SARS-CoV-2 kit.
  Serum was also tested by ELISA with the SARS-CoV-2 (IgG) ELISA Kit (EuroIm-mun, France).
  These ELISA and ECLIA tests were carried out in the medical biology laboratory of the Institut Bergonié.
  Serological immune status to a previous infection by the SARS-CoV-2 virus was evaluated for each patient and defined as :
  * Positive in case of positive ELISA test AND/OR positive ECLIA test
  * Negative otherwise
Time Frame: Time 0 (Inclusion)
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-SERO-COV
Number analyzed (Participants) | 517
Participants | 18

2. Secondary Outcome: Rate of Positive Serological Immune Status to a Previous Infection by the SARS-CoV-2 Virus at 3 Months
Description: as for outcome 1
Time Frame: 3 months
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion and at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-SERO-COV
Number analyzed (Participants) | 500
Participants | 31

3. Secondary Outcome: Rate of Positive Serological Immune Status to a Previous Infection by the SARS-CoV-2 Virus at 12 Months
Description: Total antibodies (IgG and IgM) directed against the N (nucleocapsid) protein of the virus were determined by ECLIA on a Cobas® 8000 (Roche Diagnostic, France) with the Elecsys Anti-SARS-CoV-2 kit.
  ECLIA test was carried out in the medical biology laboratory of the Institut Bergonié.
  Serological immune status to a previous infection by the SARS-CoV-2 virus was evaluated for each patients and defined as :
  * Positive in case of positive ECLIA test
  * Negative otherwise
Time Frame: 12 months
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion, 3 months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-SERO-COV
Number analyzed (Participants) | 462
Participants | 46

4. Secondary Outcome: Number of Health Care Workers With Active COVID-19 Infection
Description: Defined by a positive result for the molecular test for the detection of the SARS-CoV-2 coronavirus genome by RT-PCR.
Time Frame: Time 0 (inclusion), 3 months, 12 months
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion (for 0 month visit) , 3 months (for 3 months visit) and 12 months (for 12 months visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-SERO-COV
Number analyzed (Participants) | 517
Participants
  0 months | 0
  3 months: number analyzed (Participants) | 500
  3 months | 0
  12 months: number analyzed (Participants) | 462
  12 months | 0

5. Secondary Outcome: Number of Health Care Workers With Symptoms of Anxiety at 0 Months (Inclusion)
Description: Generalized Anxiety Disorder (GAD-7) self-questionnaire, whose score varies from 0 (no anxiety) to 21 (severe anxiety).
  Following the recommended threshold, generalized anxiety is estimated from 10 points.
Time Frame: Time 0 (inclusion)
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion and who signed informed consent form for the optional study and completed the GAD-7 at inclusion
Measure: Count of Participants; unit: Participants
Groups:
- PRO-SERO-COV (Optionnal Study): Blood sample and self-administered questionnaire
  PRO-SERO-COV: At inclusion, 3 months and 12 months :
  * blood sample (2 x 5ml)
  * self-administered questionnaire
  Informed consent form signed for the optional study
Arm/Group | PRO-SERO-COV (Optionnal Study)
Number analyzed (Participants) | 460
Participants | 36

6. Secondary Outcome: Number of Health Care Workers With Symptoms of Anxiety at 3 Months
Description: as for outcome 5
Time Frame: 3 months
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion and who signed informed consent form for the optional study and completed the GAD-7 at 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-SERO-COV (Optionnal Study)
Number analyzed (Participants) | 442
Participants | 49

7. Secondary Outcome: Number of Health Care Workers With Symptoms of Anxiety at 12 Months
Description: as for outcome 5
Time Frame: 12 months
Population: Eligible participant who completed the self-administered questionnaire and had blood sample available at inclusion and who signed informed consent form for the optional study and completed the GAD-7 at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-SERO-COV (Optionnal Study)
Number analyzed (Participants) | 413
Participants | 30

ADVERSE EVENTS:
Time Frame: As this study is an observational study, adverse events and serious adverse events were not collected.
Arm/Group | PRO-SERO-COV
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04426006/Prot_SAP_001.pdf